CLINICAL TRIAL: NCT05882591
Title: Posteromedial Tibiofemoral Incongruence (PMTFI) Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Artromedical Konrad Malinowski Clinic (Other)
Responsible Party: Principal Investigator, Konrad Malinowski MD, Konrad Malinowski MD, Director of Artromedical Konrad Malinowski Clinic and Principal Investigator, Artromedical Konrad Malinowski Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-pro-ar-2023
Record Dates: First submitted 2023-05-20; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Meniscus Disorder; Meniscus; Degeneration; Meniscus Tear; Meniscus Lesion

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main arm of the study (Experimental): Posteromedial Tibiofemoral Incongruence (PMTFI) Treatment by the means of published technique (reference nr 1).
  Interventions: Procedure: Posteromedial Tibiofemoral Incongruence (PMTFI) Treatment by the means of published technique (reference nr 1).

INTERVENTIONS:
Procedure: Posteromedial Tibiofemoral Incongruence (PMTFI) Treatment by the means of published technique (reference nr 1). — Posteromedial Tibiofemoral Incongruence (PMTFI) Treatment by the means of published technique (reference nr 1).

SUMMARY:
The aim of this study is to assess outcomes of Posteromedial Tibiofemoral Incongruence (PMTFI) Treatment

DETAILED DESCRIPTION:
The aim of this study is to assess outcomes of Posteromedial Tibiofemoral Incongruence (PMTFI) Treatment by the means of published technique (reference nr 1).

A decrease in the posterior curvature of the femoral metaphysis close to the medial femoral condyle is one of the anatomical alterations that can be seen within the knee joint. When the knee is fully flexed, this curve is typically concave enough to accommodate the posterior horn of the medial meniscus (PHMM). Similar to cam incongruence in the hip joint, a decrease in curvature may cause posteromedial tibiofemoral incongruence, a condition marked by compression of the PHMM in complete knee flexion. If deep knee flexion occurs, clinical symptoms may appear, and PHMM degeneration may be shown to worsen over time. Surgery may be recommended for patients for whom activity modification and conservative therapy have failed. Our team proposed an arthroscopic procedure that allows for the least amount of correction that is still necessary while also providing final intraoperative confirmation of the clinical need to repair posteromedial tibiofemoral incongruence.

ELIGIBILITY:
Inclusion Criteria:

* Pain, snapping or discomfort in posterior part of the knee in deep knee flexion during squat
* Reduced concavity of the femoral metaphysis proximal to the medial femoral condyle confirmed on MRI
* Impingement of posterior horn of medial meniscus with the metaphysis of femur during full knee flexion confirmed arthroscopically

Exclusion Criteria:

* Active knee inflammation
* Chondral injuries ICRS 3-4
* Extraarticular reasons of pain, snapping or discomfort in posterior part of the knee in deep knee flexion during squat
* Cyst or avascular changes within the femoral metaphysis adjacent to the planned localization of the procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of pain in full knee flexion | At the 12 month of the follow-up
  Presence of pain in full knee flexion - deep squat: pain yes/no
Presence of pain in full knee flexion | At the 24 month of the follow-up
  Presence of pain in full knee flexion - deep squat: pain yes/no

SECONDARY OUTCOMES:
The functional assessment with the The International Knee Documentation Committee Questionnaire (IKDC) | At the 12 month of the follow-up
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the The International Knee Documentation Committee Questionnaire (IKDC) | At the 24 month of the follow-up
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score (KOOS) | At the 12 month of the follow-up.
  Min of 0 max of 100 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score (KOOS) | At the 24 month of the follow-up.
  Min of 0 max of 100 points, higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Malinowski, MD PhD, Principal Investigator — Artromedical Orthopaedic Clinic, Bełchatów, Poland
Locations (1):
- Artromedical Orthopaedic Clinic, Bełchatów, Łódź Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Malinowski K, Kozlak M, Mostowy M, LaPrade RF, Ebisz M, Pekala PA. Cam Impingement of the Knee: Arthroscopic Correction of Posteromedial Tibiofemoral Incongruence. Arthrosc Tech. 2022 May 11;11(6):e951-e957. doi: 10.1016/j.eats.2022.01.015. eCollection 2022 Jun. PMID 35782837
- [Result] Suganuma J, Mochizuki R, Yamaguchi K, Inoue Y, Yamabe E, Ueda Y, Fujinaka T. Cam impingement of the posterior femoral condyle in medial meniscal tears. Arthroscopy. 2010 Feb;26(2):173-83. doi: 10.1016/j.arthro.2009.11.002. PMID 20141980
- [Result] Suganuma J. Lack of posteromedial tibiofemoral congruence at full flexion as a causative factor in isolated medial meniscal tears. J Orthop Sci. 2002;7(2):217-25. doi: 10.1007/s007760200036. PMID 11956982